CLINICAL TRIAL: NCT03918304
Title: Open Label, Multicenter, Real World Treatment Study of Single Agent Tagrisso; KOREA PLUS Study (Korea Osimertinib Real World Evidence Study to Assess Safety and Efficacy - PLUS).
Brief Title: Korea Osimertinib Real World Evidence Study to Assess Safety and Efficacy - PLUS
Acronym: KOREA-PLUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161R00005
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
This is a local, prospective, non-interventional, regulatory postmarketing surveillance study. The objectives of this study are to assess the safety and efficacy of single agent Tagrisso (Osimertinib, hereinafter "the study drug") in a real world setting according to the approved label in Korea.

DETAILED DESCRIPTION:
* Primary objective: To assess safety of the Tagrisso for patients with NSCLC treated with Tagrisso under the approved indication in Korea
* Secondary objective: To assess efficacy of the Tagrisso for patients with NSCLC treated with Tagrisso under the approved indication in Korea.

ELIGIBILITY:
* Inclusion Criteria:

  1. Eligible for, or on active study drug treatment according to the approved prescribing information;
* The first-line treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) whose tumours have epidermal growth factor receptor (EGFR) exon 19 deletions or exon 21 (L858R) substitution mutations
* Treatment of patients with locally advanced or metastatic EGFR T790M mutation-positive NSCLC who have been previously treated with EGFR TKI therapy
* The adjuvant treatment after complete tumour resection in patients with non-small cell lung cancer (NSCLC) whose tumours have epidermal growth factor receptor (EGFR) exon 19 deletions or exon 21 (L858R) substitution mutations 2. Provision of signed and dated written informed consent by the patient or legally acceptable representative
* Exclusion Criteria:

  1. History of hypersensitivity to the active substance or to any of the excipients of this drug
  2. Pregnancy and/or breast feeding
  3. Current participation in any interventional trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: On active study drug treatment according to the approved label
Sampling Method: Non-Probability Sample
Enrollment: 923 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of patients with at least one event of adverse events (AEs), serious adverse events (SAEs) and AEs of special interest (AESI) | For about 1 year since the first dose of the study drug
Severity of (S)AEs according to CTCAE | For about 1 year since the first dose of the study drug

SECONDARY OUTCOMES:
ORR (Objective response rate), if available | For about 1 year since the first dose of the study drug
PFS (Progression free survival) , if available | For about 1 year since the first dose of the study drug
DFS (Disease free survival), if available | For about 1 year since the first dose of the study drug

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Research Site, Busan
  - Research Site, Chungcheongbuk-do
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gangwon State
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Jeollabuk-do
  - Research Site, Jeollanam-do
  - Research Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/DisclosureYes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D5161R00005_Study Report Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161R00005&attachmentIdentifier=6e709bb8-f71b-43cd-8cc6-0b9f3e5bd47b&fileName=D5161R00005_Study_Report_Synopsis_redacted.pdf&versionIdentifier=